CLINICAL TRIAL: NCT04358185
Title: A Phase Ib Study of Itacitinib, a JAK1 Inhibitor, in Advanced Hepatocellular Carcinoma
Brief Title: Itacitinib in Advanced Hepatocellular Carcinoma
Acronym: JAKaL
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Imperial College London (Other)
Collaborators: Incyte Biosciences UK Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 237279; 2017-004437-81 (EudraCT Number)
Record Dates: First submitted 2020-04-17; First posted 2020-04-24 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Advanced Hepatocellular Carcinoma
MeSH Terms: interventions — itacitinib; INCB039110

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Itacitinib (Experimental): Itacitinib (INCB039110) - novel and small molecule selective inhibitor of JAK1
  Interventions: Drug: Itacitinib (INCB039110)

INTERVENTIONS:
Drug: Itacitinib (INCB039110) — Novel and small molecule selective inhibitor of JAK1

SUMMARY:
This research will assess the effects of Itacitinib as a second line treatment for patients with advanced inflammatory hepatocellular carcinoma (HCC), a type of liver cancer. Itacinib is a protein inhibitor of the tyrosine kinase, JAK1, which is believed to enable cancer cells to metastasise to other parts of the body.

DETAILED DESCRIPTION:
JAKaL is a single arm phase Ib study evaluating the effect of Itacitinib in 25 patients with advanced HCC.

Many patients diagnosed with HCC will have advanced disease where only palliative care is offered to them, this could account for the relatively low reported 5-year survival rate of approximately 10%. There are a number of epidemiological and pre-clinical studies that have investigated the role of chronic inflammatory conditions in the development of HCC and these provide evidence that inflammation promotes malignant transformation. The production of tumour-promoting cytokines by inflammatory cells can activate transcription factors, such as STAT3 via the JAK/STAT pathway in premalignant cells. STAT3, once activated, can cause the expression of further genes necessary for cell activation, localisation, survival and proliferation. Inhibition of JAK could therefore be a way of directly affecting malignant cell proliferation, as STAT3 in most malignancies are persistently phosphorylated and thereby stimulated to carry out its function; to sustain cell proliferation and block apoptosis.

For reference, STAT3 is a member of the STAT protein family and is switched on, via phosphorylation, by receptor-associated Janus kinases (JAK), a type of tyrosine kinase, and together they form homo-/heterodimers that translocate to the cell nucleus and act as transcription activators. STAT3 mediates the expression of a variety of genes and therefore is integral to many cellular processes, as mentioned above, such as cell growth and apoptosis, and thus they can promote oncogenesis by being over-active in the different signalling pathways it is involved in.

Itacitinib has not yet been approved by the U.S. Food and Drug Administration (FDA) for any clinical indication but has been developed as potential treatments for myelofibrosis (MF), rheumatoid arthritis (RA), psoriasis, graft-versus-host disease (GVHD), B cell malignancies and solid tumours like HCC. It is a small molecule selective inhibitor of JAK1 thereby preventing its phosphorylation of STAT proteins, particularly STAT3, resulting in a decrease in the expression of genes responsible for cell activation, localisation, survival and proliferation

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 or over
2. Diagnosis of hepatocellular carcinoma. If primary diagnosis of HCC: diagnosis based on the following criteria:

   * cyto-histological criteria, OR
   * radiological criteria: Focal lesion >1 cm with arterial hypervascularization in 2 coincident imaging techniques (CT, MRI, or US), OR
   * combined criteria: one imaging technique showing a focal lesion 1-2 cm with arterial hypervascularization AND AFP levels >400 ng/mL, OR
   * combined criteria: one imaging technique showing a focal lesion >2 cm with arterial hypervascularization AND AFP levels >200 ng/mL
3. Child-Pugh A and B up to 7 points (in patients receiving anticoagulant therapy; Child-Pugh score up to 5 points; INR category not regarded for calculation of the Child-Pugh score)
4. Progression or intolerance to first line therapy - N.B: Date of patients last dose of therapy must be more than 28 days before enrolment into this study.
5. ECOG Performance status 0, 1 or 2.
6. Adequate organ function as defined by:

   * Adequate hematologic function (ANC 1.0x109/l, platelet count 50x109/l, and hemoglobin 9g/dl).
   * Serum creatinine concentration < 1.5 times the upper limit of normal (ULN) and/or creatinine clearance >60 ml/min
   * Bilirubin level < 1.5 X ULN
   * PT-INR/PTT<1.5 x ULN
7. For women of child-bearing potential (defined as women who have not undergone surgical sterilization with a hysterectomy, and/or bilateral oophorectomy, and are not postmenopausal, defined as ≥12 months of amenorrhea) must have a negative serum pregnancy test within 14 days prior to the first study drug administration Effective contraception must be used throughout the duration of the study and up to 30 days following the last dose of the investigational medicinal product (IMP). Effective forms of contraception include complete abstinence from sexual intercourse, double barrier methods (condom with spermicide in conjunction with use of an intrauterine device or condom with spermicide in conjunction with use of a diaphragm), birth control patch or vaginal ring, oral, injectable, or implanted contraceptives and surgical sterilization (tubal ligation or vasectomy). Sperm and ova donation are prohibited during the duration of the study and 30days after the last dose. 8. Written informed consent prior to initiation of any study procedures and willing and able to comply with the study schedule

Exclusion Criteria:

1. Previous treatment with:

   * Study medication, any other JAK1 inhibitor and/or known hypersensitivity to the study medication
   * An investigational agent within 28 days prior to start of study treatment
2. Serious concurrent medical or psychiatric illness, including serious active infection
3. Uncontrolled ascites
4. Uncontrolled hypertension
5. History of organ transplant (including prior liver transplant)
6. Diagnosis of HIV, congenital immune defect, any immunosuppressive therapy for autoimmune disease or inflammatory bowel disease
7. Patients with active or latent tuberculosis
8. Patients with active hepatitis C or active hepatitis B that requires treatment
9. Patients who have received a live vaccine 30 days or fewer prior to enrolment as well as patients who intend to receive live vaccination during study participation or for three months after last dose administration

8. Patients who have a history of unprovoked venous thromboembolism (VTE) prior to the diagnosis of malignancy 9. Pregnant or breast feeding women Other clinically significant co-morbidities that could compromise the subject's participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of Itacitinib in patients with HCC: adverse events | Throughout study completion, up to 1 year
  Assessment of adverse events relating to experimental drug intake according to the Common Terminology Criteria for Adverse Events (CTCAE) V4.03
To assess efficacy of Itacitinib by overall response rate: objective response rate (ORR) | Throughout study completion, up to 1 year
  Measure objective response rate (ORR) as complete response, partial response, stable disease or progressive disease at 8 weeks post treatment according to RECIST criteria (mRECIST) V1.1

SECONDARY OUTCOMES:
Efficacy of Itacitinib by progression free survival | Throughout study completion, up to 1 year
  Progression free survival (PFS), defined as time from study entry to first evidence of disease progression assessed by mRECIST v1.1 or death due to any cause
Efficacy of Itacitinib by overall survival | Throughout study completion, up to 1 year
  Overall survival (OS), defined as time from study entry to death due to any cause

OTHER OUTCOMES:
Presence of predefined JAK1 mutations in tumour tissue | Throughout study completion, up to 1 year
  Assessment of presence of predefined JAK1 mutations in tumour tissue
Translational studies | Throughout study completion, up to 1 year
  Assessment of presence of predefined JAK1 mutations in ctDNA
Translational studies 2 | Throughout study completion, up to 1 year
  Correlation of changes in proinflammatory cytokines (multiplex bead array) with treatment response (mRECIST)
Correlation of JAK1 mutations with treatment | Throughout study completion, up to 1 year
  Using mRECIST to find the correlation between the presence of predefined JAK1 mutations in tumour tissue with treatment outcome

CONTACTS AND LOCATIONS:
Overall Officials: Rohini Sharma, MD, Principal Investigator — Senior Lecturer Medical Oncology and Clinical Pharmacology
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Troiani A, Martinez M, Ward C, Benartzi CW, Pinato DJ, Sharma R. Safety and efficacy of itacitinib, a selective JAK1 inhibitor, in advanced hepatocellular cancer: Phase 1b trial (JAKAL). Future Oncol. 2024;20(36):2839-2847. doi: 10.1080/14796694.2024.2396795. Epub 2024 Sep 16. PMID 39283290